CLINICAL TRIAL: NCT02376595
Title: Pharmacokinetic and Pharmacodynamic of Rocuronium Bromide Measured in Adductor Pollicis and Masseter Muscles.
Brief Title: Pharmacokinetic and Pharmacodynamic of Rocuronium
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 12-003
Record Dates: First submitted 2015-02-12; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Neuromuscular Blockade
Keywords: Rocuronium; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rocuronium Bromide: Rocuronium 0,3 mg/kg administered in less than five seconds, followed by a saline bolus.
  Interventions: Drug: Rocuronium Bromide

INTERVENTIONS:
Drug: Rocuronium Bromide — Rocuronium 0,3 mg/kg in less than five seconds, followed by a saline bolus.
  Other Names: Rocuronium Bromide Fresenius Kabi

SUMMARY:
The purpose of this study is characterize the dose-effect relationship of rocuronium bromide at the adductor pollicis and masseter muscles using an pharmacokinetic-pharmacodynamic (PKPD) model. The hypothesis is that masseter muscle has a greater sensitivity to the neuromuscular blockers (rocuronium), faster onset and slower recovery profile than the adductor pollicis muscle.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery under general anesthesia.

Exclusion Criteria:

* Pregnancy.
* Body mass index (BMI) >25 kg/m2.
* Anticipated difficult airway.
* Surgery associated with great volume loss.
* Presence of any neuromuscular, hepatic, renal, cardiac or respiratory disease.
* Previous history of neuromuscular blockade allergy, and/or administration of drugs known to interfere with neuromuscular blockade

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 ASA I-II patients, aged 18-65 years, scheduled for elective surgery under general anesthesia, were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
strength measuring 2 acceleromyograph. One Placed at the masseter muscle and the other one at the adductor pollicis muscle. | 60 minutes
Measure blood concentrations after administration rocuronium | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Luis I Cortinez, MD, Study Chair — Ponticia Universidad Católica

REFERENCES:
- [Background] Plaud B, Proost JH, Wierda JM, Barre J, Debaene B, Meistelman C. Pharmacokinetics and pharmacodynamics of rocuronium at the vocal cords and the adductor pollicis in humans. Clin Pharmacol Ther. 1995 Aug;58(2):185-91. doi: 10.1016/0009-9236(95)90196-5. PMID 7648768
- [Background] Donati F, Meistelman C, Plaud B. Vecuronium neuromuscular blockade at the adductor muscles of the larynx and adductor pollicis. Anesthesiology. 1991 May;74(5):833-7. doi: 10.1097/00000542-199105000-00006. PMID 1673592
- [Background] Saitoh Y, Oshima T, Nakata Y. Acceleromyographic monitoring of neuromuscular block over the orbicularis oris muscle in anesthetized patients receiving vecuronium. J Clin Anesth. 2010 Aug;22(5):318-23. doi: 10.1016/j.jclinane.2009.09.004. PMID 20650376
- [Background] Kitajima O, Suzuki T, Fukano N, Saeki S, Ogawa S, Noda Y. Onset of rocuronium-induced neuromuscular block evaluated subjectively and accerelomyographically at the masseter muscle. J Anesth. 2011 Jun;25(3):376-9. doi: 10.1007/s00540-011-1129-0. Epub 2011 Apr 12. PMID 21484503
- [Background] Cantineau JP, Porte F, d'Honneur G, Duvaldestin P. Neuromuscular effects of rocuronium on the diaphragm and adductor pollicis muscles in anesthetized patients. Anesthesiology. 1994 Sep;81(3):585-90. doi: 10.1097/00000542-199409000-00010. PMID 8092503
- [Background] Ibebunjo C, Srikant CB, Donati F. Morphological correlates of the differential responses of muscles to vecuronium. Br J Anaesth. 1999 Aug;83(2):284-91. doi: 10.1093/bja/83.2.284. PMID 10618945
- [Background] Smith CE, Donati F, Bevan DR. Differential effects of pancuronium on masseter and adductor pollicis muscles in humans. Anesthesiology. 1989 Jul;71(1):57-61. doi: 10.1097/00000542-198907000-00011. PMID 2751140
- [Background] Zhang L, Beal SL, Sheiner LB. Simultaneous vs. sequential analysis for population PK/PD data I: best-case performance. J Pharmacokinet Pharmacodyn. 2003 Dec;30(6):387-404. doi: 10.1023/b:jopa.0000012998.04442.1f. PMID 15000421
- [Background] Schnider TW, Minto CF, Gambus PL, Andresen C, Goodale DB, Shafer SL, Youngs EJ. The influence of method of administration and covariates on the pharmacokinetics of propofol in adult volunteers. Anesthesiology. 1998 May;88(5):1170-82. doi: 10.1097/00000542-199805000-00006. PMID 9605675
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Viby-Mogensen J, Ostergaard D, Donati F, Fisher D, Hunter J, Kampmann JP, Kopman A, Proost JH, Rasmussen SN, Skovgaard LT, Varin F, Wright PM. Pharmacokinetic studies of neuromuscular blocking agents: good clinical research practice (GCRP). Acta Anaesthesiol Scand. 2000 Nov;44(10):1169-90. doi: 10.1034/j.1399-6576.2000.441002.x. PMID 11065197
- [Background] Cho HE, Park MJ, Kim SC, Hong RS, Moon DC, Ahn SY. Analysis of rocuronium in human whole blood and tissues using liquid chromatography-tandem mass spectrometry. J Chromatogr Sci. 2013 Apr;51(4):297-301. doi: 10.1093/chromsci/bms252. Epub 2013 Feb 1. PMID 23377654
- [Background] Zhang L, Beal SL, Sheinerz LB. Simultaneous vs. sequential analysis for population PK/PD data II: robustness of methods. J Pharmacokinet Pharmacodyn. 2003 Dec;30(6):405-16. doi: 10.1023/b:jopa.0000012999.36063.4e. PMID 15000422
- [Background] Sheiner LB, Stanski DR, Vozeh S, Miller RD, Ham J. Simultaneous modeling of pharmacokinetics and pharmacodynamics: application to d-tubocurarine. Clin Pharmacol Ther. 1979 Mar;25(3):358-71. doi: 10.1002/cpt1979253358. PMID 761446
- [Background] Dragne A, Varin F, Plaud B, Donati F. Rocuronium pharmacokinetic-pharmacodynamic relationship under stable propofol or isoflurane anesthesia. Can J Anaesth. 2002 Apr;49(4):353-60. doi: 10.1007/BF03017322. PMID 11927473
- [Background] Kuipers JA, Boer F, Olofsen E, Bovill JG, Burm AG. Recirculatory pharmacokinetics and pharmacodynamics of rocuronium in patients: the influence of cardiac output. Anesthesiology. 2001 Jan;94(1):47-55. doi: 10.1097/00000542-200101000-00012. PMID 11135721
- [Background] De Mey JC, De Baerdemaeker L, De Laat M, Rolly G. The onset of neuromuscular block at the masseter muscle as a predictor of optimal intubating conditions with rocuronium. Eur J Anaesthesiol. 1999 Jun;16(6):387-9. doi: 10.1046/j.1365-2346.1999.00503.x. PMID 10434167
- [Background] Nakamura Y, Torisu T, Noguchi K, Fujii H. Changes in masseter muscle blood flow during voluntary isometric contraction in humans. J Oral Rehabil. 2005 Aug;32(8):545-51. doi: 10.1111/j.1365-2842.2005.01461.x. PMID 16011632
- [Background] Abdulatif M, el-Sanabary M. Blood flow and mivacurium-induced neuromuscular block at the orbicularis oculi and adductor pollicis muscles. Br J Anaesth. 1997 Jul;79(1):24-8. doi: 10.1093/bja/79.1.24. PMID 9301384